CLINICAL TRIAL: NCT05335616
Title: Behavioral Change Simulation Experiment Regarding Dentists' Repair Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Göttingen (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Philipp Kanzow, PD Dr. med. dent., Dr. rer. medic., Senior Dental Practitioner, University Medical Center Goettingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Repair-SimulationExperiment; 22/4/22 (Other: Local Ethics Commission)
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Behavior
Keywords: decision-making; repair behavior; questionnaire
MeSH Terms: conditions — Behavior | interventions — Guidelines as Topic

STUDY DESIGN:
Intervention Model Description: Either of two potential interventions is delivered as written instruction to the participants
Masking Description: Intervention will be delivered in a separate, sealed envelope. Thereby, participants are blinded for the intervention when baseline data will be gathered (i.e. by filling out the first questionnaire).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention "Guideline" (Experimental): Participants are given written information (a hypothetical new guideline).
  Interventions: Other: Guideline
- Intervention "Treatment fee item" (Experimental): Participants are given written information about a hypothetical new treatment fee item.
  Interventions: Other: Treatment fee item

INTERVENTIONS:
Other: Guideline — Hypothetical guideline regarding the indications and treatment steps involved in dental restoration repair.
  Arms: Intervention "Guideline"
Other: Treatment fee item — Arrangement of a hypothetical treatment fee item which can be charged in addition to the actual repair restoration.
  Arms: Intervention "Treatment fee item"

SUMMARY:
The aim of the present study is to determine the effect of two potential interventions on dentists' behavior regarding the repair of partially defective dental restorations.

DETAILED DESCRIPTION:
Two potential interventions are delivered as written instructions to the participants. Dentists are asked to indicate their treatment preference for two given clinical scenarios (consisting of case vignettes, clinical photos, and radiographs) in two questionnaires prior (baseline data) and after receiving the intervention. Based on these data, the simulated behavior change (i.e. to repair or not to repair) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* General dentists, working in Germany and being listed in an address databse (www.adressdiscount.de)

Exclusion Criteria:

* Dentists who are not listed in the above-mentioned database
* Dentists who have previously declined to participate in future research from our department.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2944 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Simulated behavior change | 10 Minutes
  Simulated behavior change, indicated by the proportion of dentists selecting repairs as their treatment preference for the given clinical scenarios.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Goettingen, Dept. of Preventive Dentistry, Periodontology and Cariology, Göttingen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kanzow P, Kanzow AF, Wiegand A, Schwendicke F. Implementation of repairs in dental practice: Randomized behavior simulation trial. J Am Dent Assoc. 2023 Jul;154(7):610-619.e11. doi: 10.1016/j.adaj.2023.04.007. Epub 2023 May 22. PMID 37212760